CLINICAL TRIAL: NCT03538119
Title: Phase III Cardiac Rehabilitation in Coronary Patients: High-intensity Interval Training or Moderate-intensity Continuous Training?
Brief Title: Comparison Between HIIT and MICT on the Phase III of Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Catarina Joaquim Gonçalves, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR_UEvora
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Patients With Coronary Artery Disease
Keywords: Cardiac Rehabilitation; High Intensity Interval Training; Moderate Intensity Continuous Training; Secondary prevention; Cardiovascular Risk Factors; Exercise-based Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training Program (Experimental): Three sessions of exercises will be performed weekly with duration of 30 min to 45 min, divided into warm up, aerobic exercise (4x4 high-intensity intervals at 85%-95%) and recovery.
  Interventions: Other: High Intensity Interval Training Program
- Moderate Intensity Continuous Training Program (Experimental): Three sessions of exercises will be performed weekly with duration of 45 min to 60 min, divided into warm up, aerobic exercise (continuous intensity at 70-75%HRpeak) and recovery.
  Interventions: Other: Moderate Intensity Continuous Training Program
- Control Group (No Intervention): Usual care. The patients will receive nutritional counseling as well as physical activity.

INTERVENTIONS:
Other: High Intensity Interval Training Program — The HIIT group performed 4 × 4-minute high-intensity intervals at 85%-95% HRpeak followed by a 1-minute recovery interval at 40% HRpeak, predicted with a supervised graded exercise test on a treadmill with the Bruce protocol. The protocol will include a warm-up of 10 minutes at low moderate intensity (50-70% of HRpeak) and a 3 to 5 minute calm return period at 50% of the HRpeak.
  The supervised sessions will take place on treadmill, 3 times a week for 6 consecutive weeks. If a session is lost, it will be recovered that week or the following week. Each session will be limited to three participants.
  Other Names: HIIT
  Arms: High Intensity Interval Training Program
Other: Moderate Intensity Continuous Training Program — The MICT protocol (usual care) consisted of a continuous bout of moderate-intensity exercise to elicit 70-75% HRpeak, rating of perceived exertion 3 to 5 (fairly light to somewhat hard), for 27.5 minutes to equate the energy expenditure with the HIIT protocol. The protocol will include a warm-up of 10 minutes at low moderate intensity (50-70% of HRpeak) and a 3 to 5 minute calm return period at 50% of the HRpeak.
  The supervised sessions will take place on treadmill, 3 times a week for 6 consecutive weeks. If a session is lost, it will be recovered that week or the following week. Each session will be limited to three participants.
  Other Names: MICT
  Arms: Moderate Intensity Continuous Training Program

SUMMARY:
The increase in the prevalence of cardiovascular diseases (CVD), directly associated with the aging of the population, is a concern for public health in Portugal. Given the high prevalence of risk factors and the increasing number of cases of CD throughout Alentejo, where there is no cardiac rehabilitation (CR) coverage, there is an urgent need for the implementation of a CR program.

CR has evolved over the past decades to multidisciplinary approaches focused on education, individualized training, modification of risk factors, and overall well-being of cardiac patients. Studies suggest that high intensity interval training (HIIT) allows greater patient benefits compared to moderate continuous training (MCT), reversal of DC and increased aerobic capacity in CR patients. This study intends to compare HIIT and MCT interventions investigating direct and indirect associations between informally performed physical activity (AF), sedentary behavior, cardiovascular fitness and quality of life (QoL) among patients enrolled in RC programs in phase III.

DETAILED DESCRIPTION:
According to WHO (1) cardiovascular diseases (CVD) are the number 1 cause of death globally: an estimated 17.5 million people died from CVD in 2012, representing 31% of all global deaths. In 2013 there were 1.9 million deaths resulting from CVD of the circulatory system in the EU-28, which was correspondent to 37.5 % of all deaths considerably higher than the second most prevalent cause of death, cancer.

In Portugal, cardiovascular diseases lead to morbidity and mortality rates, which makes evident the importance in the Public Health scenario and the need to implement measures aimed at primary and secondary prevention. In 2004, cardiovascular diseases signify 39% of all causes of death, since then a reduction in these values has been recorded and, according to more recent data (2013), the values are around 29.5%.

As these pathologies are associated, among other causes, with aging, the Alentejo emerges as one of the regions where the prevalence of these pathologies is greater. In fact, since Alentejo is the oldest region, it becomes an authentic Living Lab. In this way, this study intends to study the effects of different types of cardiac rehabilitation (CR) programs, emphasizing in particular the use of a high intensity interval program that we will compare with a traditional program.

For the program will be recruited patients who have been admitted in the Cardiology Services at Espírito Santo Hospital in Évora. Participants of both sexes will be included, between 18 and 80 years of age, meeting the criteria for low or moderate risk, class B for participation and exercise supervision, absence of signs/symptoms after cardiac surgery, with a left ventricular ejection fraction greater than 40%, according to the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation.

Those who meet the inclusion criteria will be evaluated in a clinical context in order to determine the capacity to integrate phase III of CR. This phase will last about 6 weeks, will be held at the Nursing School located at the Espírito Santo Hospital.

The sessions will be supervised and will take place on a cycloergometer and treadmill, 3 times a week for 6 consecutive weeks. If a session is lost, it will be recovered that week or the following week. Each session will be limited to three participants.

The HIIT protocol will consist of four four-minute intervals at high intensity, stimulating 85-95% of peak-FC followed by active recovery at 70% peak-FC for a total of 20 minutes. The MCT protocol consists of continuously exerting moderate intensity, causing a peak-FC 70-75% for 27.5 minutes to equal the energy expenditure of the HIIT protocol. Both protocols will include a warm-up of 10 minutes at low moderate intensity (50-70% of peak-FC) and a 3 to 5 minute calm return period was performed at 50% of peak-FC.

During the intervention, the workload, FC and the subjective effort perception scale (EPE - Borg) will be recorded throughout each session, every minute for the HIIT training and all other minutes for the MTC. During the intervention the load will be adjusted to obtain the target FC.

After the exercise session, participants will complete 1 of 18 items of the Physical Activity and Pleasure Scale (PACES) on a weekly basis in which subjects rate their appreciation for the exercise of that week on a seven-point scale.

In the same period, the usual medical recommendations for cardiac rehabilitation through exercise will be provided to the Control Groups (phase III).

When subjects complete phase III CR, they will be given guidelines on exercise and nutrition. The intention is that participants after the program have adopted a healthy lifestyle, where the practice of physical exercise is a reality. The intention is also to verify if participation in one of the different exercise programs that have been implemented, in phase III of CR, can possibly provide better results both in maintaining good life habits and also in reducing the time in the sedentary activities, the "Active Couch Potato" phenomenon. More than solving a health problem at a certain stage of a subject's life, it is intended to consolidate healthy habits of life.

In order to verify which type of program allows to modify the habits of life towards the increase of the practice of physical activity, as well as the maintenance of these habits, we will carry out a follow-up at 6 months and one year after the beginning of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* low-moderate risk for physical exercise, with the following pathologies / conditions:
* stable coronary disease;
* after acute myocardial infarction;
* after coronary angioplasty;
* after cardiac surgery (coronary revascularization or valve surgery);
* stable chronic heart failure in class I-II of the New York Heart Association;
* acceptance of the informed consent assumptions of CR programs;
* must not have participated in physical exercise programs in the 3 months preceding the referral;
* should not have more than one hour of vigorous physical activity per week according to the International Physical Activity Questionnaire.

Exclusion Criteria:

* presenting symptoms of heart failure of class III and IV according to the New York Heart Association (or documented signs and symptoms of chronic heart failure with ejection fraction >45%);
* uncontrolled arrhythmias;
* severe chronic obstructive pulmonary disease;
* uncontrolled hypertension;
* symptomatic peripheral arterial disease; unstable angina;
* uncontrolled diabetes;
* inability to perform a maximum VO2 test;
* locomotion exclusively dependent on mechanical means.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline between and within groups comparison in Blood Pressure Profile | 0 weeks, 6 weeks, 6 months and 12 months
  Systolic and diastolic blood pressure, in mmHg, and Basal Heart Rate, in heart beats per minute, to assess blood pressure profile.
Change from Baseline between and within groups comparison in Lipid Profile | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with blood tests to assess fasting triglyceride levels (mg/dL), total cholesterol (mg/dL), HDL cholesterol (mg/dL), LDL cholesterol (mg/dL), insulin (mg/dL) and glucose (mg/dL)
Change from Baseline between and within groups comparison in Body Composition | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the Dual-energy X-ray Absorptiometry to assess body fat mass (%) and body lean mass (%)
Change from Baseline between and within groups comparison in Aerobic Capacity | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the 6 Minute Walking Test, in meters, to assess aerobic capacity
Change from Baseline between and within groups comparison in Muscle Strength | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the Biodex (Peak Torque) to assess lower body muscle strength
Change from Baseline between and within groups comparison in Physical Activity Levels | 0 weeks, 6 weeks, 6 months and 12 months
  Patients were asked to wear a triaxial accelerometer (ActiGraph GT3X) on their hip placed anterior to the right iliac crest for 7 consecutive days during waking except when bathing or swimming. Acceleration data from the 3 planes were processed with ActiGraph software (ActiLife, version 6) using 15-s epochs (raw data recorded at 30 Hz) and the standard filter and were integrated into a vector magnitude count by taking the square root of the sum of squared axes (vertical, anterior-posterior, and medial-lateral).

SECONDARY OUTCOMES:
Change from Baseline between and within groups comparison in Health-related Quality of Life | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the Short Form Health Survey 36 (SF-36V2) questionnaire, total score, to assess health-related quality of life. The questionnaire consisted of the rating scale, Short Form 36 (SF-36 Quality Metric, Lincoln, Rhode Island, USA), with eight domains: physical functioning, role-physical, role-emotional, social functioning, mental health, vitality, bodily pain and general health. This instrument addresses health concepts from the patient's perspective and the scores range from 0 (worst) to 100 (best).
Change from Baseline between and within groups comparison in Anxiety and Depression | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the Hospital Anxiety and Depression Scale (HADS) questionnaire, total score, to assess health-related anxiety and depression levels. The total HADS score ranged between 0-42 with 0-14 being considered as low, 15-28 considered as moderate, and 29-42 being considered as high. For each subscale (anxiety and depression subscales), the scores ranged between 0 to 21, where 0-7 was considered low, 8-14 being moderate, while 15-21 was considered high.
Change from Baseline between and within groups comparison in Bone Composition | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with Dual-energy X-ray Absorptiometry to assess bone mineral density (g/cm2)
Change from Baseline between and within groups comparison in Sleep Quality | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the Actigraph accelerometers, in Actigraph wGT3X-BT, during 7 days of a normal week, covering 5 days weeks and 2 days of weekend to analyze sleep quality. patients were asked to wear a triaxial accelerometer (ActiGraph GT3X) on their hip placed anterior to the right iliac crest for 7 consecutive days during sleeping hours. Acceleration data from the 3 planes were processed with ActiGraph software (ActiLife, version 6) using 15-s epochs (raw data recorded at 30 Hz) and the standard filter and were integrated into a vector magnitude count by taking the square root of the sum of squared axes (vertical, anterior-posterior, and medial-lateral).

OTHER OUTCOMES:
Change from Baseline between and within groups comparison in Aerobic Capacity | 0 weeks, 6 weeks, 6 months and 12 months
  Evaluated with the Balke treadmill protocol to assess aerobic capacity response (ml.kg 1.min 1)
Change from Baseline between and within groups comparison in the Perceived Exertion during intervention | 0 weeks, 6 weeks, 6 months and 12 months
  The Borg Scale is a 10-point scale ranging from 0 to 10 with anchors ranging from ''No exertion at all'' (0) to ''Maximal exertion''. Patients were asked to rate their exertion before (pre-exercise), minute to minute of exercise, and post-exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Gonçalves, Principal Investigator — University of Évora
Locations (1):
- Catarina Gonçalves, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung ME, Bourne JE, Little JP. Where does HIT fit? An examination of the affective response to high-intensity intervals in comparison to continuous moderate- and continuous vigorous-intensity exercise in the exercise intensity-affect continuum. PLoS One. 2014 Dec 8;9(12):e114541. doi: 10.1371/journal.pone.0114541. eCollection 2014. PMID 25486273
- [Background] Heisz JJ, Tejada MG, Paolucci EM, Muir C. Enjoyment for High-Intensity Interval Exercise Increases during the First Six Weeks of Training: Implications for Promoting Exercise Adherence in Sedentary Adults. PLoS One. 2016 Dec 14;11(12):e0168534. doi: 10.1371/journal.pone.0168534. eCollection 2016. PMID 27973594
- [Background] Bartlett JD, Close GL, MacLaren DP, Gregson W, Drust B, Morton JP. High-intensity interval running is perceived to be more enjoyable than moderate-intensity continuous exercise: implications for exercise adherence. J Sports Sci. 2011 Mar;29(6):547-53. doi: 10.1080/02640414.2010.545427. PMID 21360405
- [Background] Little JP, Jung ME, Wright AE, Wright W, Manders RJ. Effects of high-intensity interval exercise versus continuous moderate-intensity exercise on postprandial glycemic control assessed by continuous glucose monitoring in obese adults. Appl Physiol Nutr Metab. 2014 Jul;39(7):835-41. doi: 10.1139/apnm-2013-0512. Epub 2014 Feb 18. PMID 24773254
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Martinez N, Kilpatrick MW, Salomon K, Jung ME, Little JP. Affective and Enjoyment Responses to High-Intensity Interval Training in Overweight-to-Obese and Insufficiently Active Adults. J Sport Exerc Psychol. 2015 Apr;37(2):138-49. doi: 10.1123/jsep.2014-0212. PMID 25996105
- [Background] Oliveira BR, Slama FA, Deslandes AC, Furtado ES, Santos TM. Continuous and high-intensity interval training: which promotes higher pleasure? PLoS One. 2013 Nov 26;8(11):e79965. doi: 10.1371/journal.pone.0079965. eCollection 2013. PMID 24302993
- [Background] Wisloff U, Ellingsen O, Kemi OJ. High-intensity interval training to maximize cardiac benefits of exercise training? Exerc Sport Sci Rev. 2009 Jul;37(3):139-46. doi: 10.1097/JES.0b013e3181aa65fc. PMID 19550205
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Derived] Goncalves C, Raimundo A, Abreu A, Pais J, Bravo J. Effects of High-Intensity Interval Training vs Moderate-Intensity Continuous Training on Body Composition and Blood Biomarkers in Coronary Artery Disease Patients: A Randomized Controlled Trial. Rev Cardiovasc Med. 2024 Mar 11;25(3):102. doi: 10.31083/j.rcm2503102. eCollection 2024 Mar. PMID 39076951
- [Derived] Goncalves C, Bravo J, Pais J, Abreu A, Raimundo A. Improving Health Outcomes in Coronary Artery Disease Patients with Short-Term Protocols of High-Intensity Interval Training and Moderate-Intensity Continuous Training: A Community-Based Randomized Controlled Trial. Cardiovasc Ther. 2023 Dec 18;2023:6297302. doi: 10.1155/2023/6297302. eCollection 2023. PMID 38146531